CLINICAL TRIAL: NCT01195064
Title: Endothelial Function Study Before Cardiovascular Surgery in COPD and/or SAS Patients
Brief Title: Endothelial Function Study Before Cardiovascular Surgery
Acronym: COPD-OSAS
Status: Terminated | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: RCB 2009-A00916-51, CHU 0921
Record Dates: First submitted 2010-06-01; First posted 2010-09-03 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Obstructive Sleep Apnea Syndrome (OSAS)
Keywords: COPD patients; OSAS patients; cardiovascular surgery; Endothelial function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urinary, blood and adipose tissue samples will be collected for measurement of different parameters of inflammation and oxidative stress.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- COPD+ OSAS- patients: Patients with chronic obstructive pulmonary disease (COPD) and without obstructive sleep apnea syndrome (OSAS), before planned cardiovascular surgery
- COPD- OSAS+ patients: Patients with obstructive sleep apnea syndrome (OSAS) and without chronic obstructive pulmonary disease (COPD), before planned cardiovascular surgery
- COPD+ OSAS+ patients: Patients with chronic obstructive pulmonary disease (COPD) and with obstructive sleep apnea syndrome (OSAS), with planned cardiovascular surgery
- COPD- OSAS- patients: Patients without chronic obstructive pulmonary disease (COPD) and without obstructive sleep apnea syndrome (OSAS), before planned cardiovascular surgery

SUMMARY:
The aim of this clinical trial is to evaluate the effect of chronic obstructive pulmonary disease (COPD) and/or obstructive sleep apnea syndrome (OSAS) on the endothelial function, before cardiovascular surgery, compared to non COPD non OSAS patients undergoing also a cardiovascular surgery, by an observational physiological study.

An interim analysis will be performed when 100 patients will be included.

DETAILED DESCRIPTION:
Secondary objectives of this clinical trial :

* To evaluate the effect of COPD and/or OSAS on the systemic inflammation, insulin-resistance and oxydative stress, in comparison with non COPD non OSAS patients.
* To evaluate the effect of COPD and/or OSAS on the inflammation and oxydative stress of the adipose tissue, in comparison with non COPD non OSAS patients.
* To validate the STOP-BANG questionnaire in patients undergoing a cardiovascular surgery

ELIGIBILITY:
Inclusion Criteria:

* Men or women between 18 and 80 years old
* Patient with planned coronary artery bypass graft surgery
* Patient with planned peripheral vascular surgery
* Patient with aortic surgery

Exclusion Criteria:

* Patient with aortic or mitral valvular replacement
* Patient with emergency peripheral valvular surgery
* Patient with emergency coronary artery bypass graft surgery
* Patient with evolutive malignancy disease
* Pregnant or lactating women
* Patient with inadvisable bronchodilator (used for functional respiratory) exploration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with chronic obstructive pulmonary disease (COPD) and/or obstructive sleep apnea syndrome (OSAS) or control patients without these pathologies, before planned cardiovascular surgery.
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2010-04; Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the percent of peripheral arterial tone (PAT) in COPD and/or OSAS patients compared to non COPD non OSAS patients. | one week before their cardiovascular surgery

SECONDARY OUTCOMES:
Evaluation of the systemic inflammation, insulin-resistance and oxidative stress occurring during COPD and/or OSAS patients compared to non COPD non OSAS patients. | one week before their cardiovascular surgery
Evaluation of adipose tissue inflammation and oxidative stress occurring during COPD and/or OSAS patients compared to non COPD non OSAS patients. | one week before their cardiovascular surgery
Polysomnography | one week before their cardiovascular surgery
Functional respiratory exploration | one week before their cardiovascular surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, MD, PhD, Principal Investigator — University Hospital of Grenoble, France
Locations (3):
- France (3):
  - University Hospital of Angers, Angers
  - Mutualist Hospital group, Grenoble
  - University Hospital of Grenoble, Grenoble

REFERENCES:
- [Background] Fabbri LM, Rabe KF. From COPD to chronic systemic inflammatory syndrome? Lancet. 2007 Sep 1;370(9589):797-9. doi: 10.1016/S0140-6736(07)61383-X. No abstract available. PMID 17765529